CLINICAL TRIAL: NCT06047275
Title: Development of Point-of-care and Wearable Sensors for Hepatitis C Diagnostics
Brief Title: HCV Microfluidic Diagnostics
Status: Completed | Type: Observational
Sponsor: University of Hull (Other)
Collaborators: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RS193 - 323660
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test: Hep C positive
- Control: Hep C negative

SUMMARY:
Hepatitis C diagnostic devices have been developed at the University of Hull to detect and quantify the Hepatitis C virus in patients' plasma and serum samples. This study aims to test the new point-of-care devices that are designed to be low cost and user-friendly.

Excess, stored, HCV patients' plasma, serum and blood samples will be supplied by the Virology laboratory (Hull University Teaching Hospital's Trust; HUTH). These samples were taken and analysed as part of patients' clinical monitoring, and are stored prior to disposal in the Virology laboratory. The proposed study will use the samples in a fully anonymised manner.

ELIGIBILITY:
Inclusion Criteria:

* Blood sample taken

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with potential Hep C
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Validation of Microfluidic device with serum and plasma | 30 minutes
  A new paper and electrochemical microfluidic device was tested with serum and plasma samples from known HCV positive samples and normal controls. The controls allowed a threshold level to be determined and all plasma and serum samples gave positive results and these were correlated with the previously acquired clinical data.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hull, Hull, United Kingdom